# MODEL INFORMED CONSENT DOCUMENT AGREEMENT TO BE IN A RESEARCH STUDY

NAME OF SPONSOR COMPANY: FORBIUS (FORMATION BIOLOGICS, CORP.

**CITY AND STATE:** Austin, Texas, USA

STUDY NAME: A Phase 1a/2a Cohort Dose Escalation Trial to Determine the

Safety, Tolerance, Maximum Tolerated Dose, and Preliminary Antineoplastic Activity of AVID100, an Anti-Human Epidermal Growth Factor Receptor (EGFR) Monoclonal Antibody Linked

to the Maytansinoid DM1, in Patients with Advanced or

Metastatic Solid Tumors of Epithelial Origin

STUDY NUMBER: AVID100-01 (Version 11; 30May2020)

Model Informed Consent (Version 5; 30May2020)

NAME OF STUDY DOCTOR: (to be completed)
TELEPHONE NUMBER(S): (to be completed)
PATIENT: (to be completed)

#### INTRODUCTION

You are being invited to take part in a research study. The doctors at <u>site</u> study the nature of cancer in an attempt to develop improved methods of diagnosis and treatment. They are conducting this study to assist Formation Biologics, Inc. (also known as Forbius, and hereafter referred to as the Sponsor) in studying an investigational drug called AVID100 (hereafter referred to as the study medication or study drug).

AVID100 is referred to as an investigational drug because it is in the early stages of development and has not been approved by any regulatory authority, which means that it is not available to be prescribed or sold. It is being tested as a possible treatment for your disease. You are being asked to take part in this study because you have a particular type of solid tumor cancer (either breast cancer, cancer of the head and neck, or lung cancer) that the study hopes to evaluate, and your disease has not responded to conventional treatment.

It is important for you to know that the doctors involved in the study have no financial interest in either Formation Biologics or the results of this study. In addition, it is important for you to know that Formation Biologics is providing the funding to cover the costs of conducting this study.

Before you decide if you want to join this study, it is important for you to know why the research is being done, how your information will be used, what the study will involve, and the possible benefits, risks, and discomforts, so that you can make an informed decision about whether you wish to participate. This process is known as "informed consent." This document that you are reading is referred to as a "consent

form" and it gives detailed information about the study, as well as how your confidentiality will be maintained. No further tests or procedures will be required of you for this study other than those that are described in this form.

Please take as much time as you need to carefully read this consent form. Some words may be new to you, and you may find some of the language difficult to understand. If so, please ask questions. The information it contains will be discussed with you. If there is anything you do not understand, or if you would like more information, please ask the study doctor or study staff. You may also discuss the study with your family, friends, and your own physician if you wish.

If you decide that you want to join this study, you will be asked to sign this consent form before having any assessments or tests performed. The study staff will give you a copy to take home with you to review prior to signing if you wish, and if you sign it, you will be given a copy of the signed version for your records. You will not be able to begin the study until you have read and signed this form.

Please know that you are free to refuse to participate in this study, and if you agree to join, you are free to leave the study at any time without having to give a reason. A decision not to take part in this study, or to withdraw at any time, will not affect your health care in any way.

#### 1. BACKGROUND AND PURPOSE OF THE STUDY

Cancer is a destructive process caused by abnormal, out of control growth of cells. Cancers (or malignancies) fall into two categories. Blood (or hematologic) cancers are the result of an abnormal growth of cells in the blood, bone marrow or lymph cells of the body. Solid tumor cancers consist of an abnormal growth of cells in other body tissues such as the lung, breast, colon, prostate, ovary, stomach, or liver. In advanced stages of disease, solid tumors may spread from the organ where they began to other organs of the body, a process called metastasis, and as a result cause far-reaching damage. Epithelial malignancies are a particular group of solid tumor cancers that come from tissues lining the external (skin) and internal (mucus membrane) surfaces of the body, and are the types of cancers this study will evaluate.

You are being invited to take part in this research study because you have an "epithelial" solid tumor cancer, one of the types to be tested in this study (either breast cancer, cancer of the head and neck, or lung cancer), and standard treatments have either failed to control your disease, you are unable to tolerate the side effects, or no effective therapy is available. Before agreeing to join this study, you should discuss with your study doctor whether all standard therapies that are available for your cancer have been tried. Once such drug to discuss, if you have a cancer of the head and neck, is cetuximab which is approved by the U.S. Food and Drug Administration (FDA) for use in patients with advanced forms of head and neck cancer after a therapy that contains a platinum-based drug has been shown not to work or not be tolerated.

As a potential drug for the treatment of cancer, AVID100, the study medication, is a combination of an antibody that is known to target the surface of certain types of cancer cells, joined by a chemical linker to a drug that is known to kill certain types of cancer cells (a cancer chemotherapy drug). As a result, AVID100 is thought to work by reaching cancer cells, and then damaging or killing them, thereby affecting how cancer cells grow and spread. This is the first study to test AVID100 in humans. AVID100 is not known to be a cure, but it is being tested to see if it can stop or control your illness.

At this point, we neither know whether the study medication will provide any benefit for cancer patients, nor do we know all of the side effects that may occur when patients receive the study medication. Studies performed with AVID100 in monkeys have shown how the drug is handled in these animals, and have provided early information about the possible side effects. These animal studies have allowed us to choose the starting dose level for studies in humans, and identify a range of higher dose levels that we believe may be safe to give to patients. Extensive research has shown that with higher doses of cancer medication there is generally a greater likelihood of patients responding to treatment. However, there is also a higher chance of side effects.

If you decide to participate, you will be monitored carefully throughout the study. At the first sign of an unacceptable side effect your doctor will decide how best to take care of you, including removing you from the study if your doctor feels this is in your best interest.

This study will be conducted in two parts, Part 1 and Part 2 (or Phase 1 and Phase 2).

- Part 1 has been completed. The main goal of Part 1 was to determine the highest dose of the study medication that can be given safely and with the least harmful side effects to patients with epithelial solid tumor cancers.
- Part 2 is ongoing. The main goals of Part 2 will be to test further the safety and effects of that highest safe dose in additional patients who have specific types of epithelial solid tumor cancers. The specific types of tumors to be tested are: 1) advanced breast cancer; 2) cancers of the head and neck; and 3) lung cancer.

You are being invited to participate in Part 2 of the trial. Your study doctor will explain the requirements of this part when he or she discusses this study with you.

#### 2. DESCRIPTION OF THE STUDY

#### What kind of study is this?

• Part 2 is an open-label study. "Open-label" means that the study doctor knows exactly what treatment is being given to each patient. The highest dose determined to be safe in Part 1 is being given to all patients in Part 2.

#### What doses of study medication will be tested, and what dose will I receive?

In Part 1 increasingly higher doses of study medication were tested in small groups of patients. Doses tested were based on a calculation of a patient's height and body weight (referred to as "body surface area"). The highest safe dose tested was the dose of 220 milligrams per meter squared per dose (220 mg/m²).

This is the dose you will receive, unless the study doctor decides a lower dose will be safer for you.

#### How will the study medication be given to me?

The study medication will be given intravenously (in the vein). Before you are given study medication, a needle will be used to insert a thin, flexible tube (catheter) into one of your veins, usually in your arm. You will receive the study medication into your vein through this flexible tube, a procedure referred to as an intravenous infusion, or an IV infusion. If you already have a catheter or a port that allows doctors to

give you medication into one of your veins, consideration will be given to using this to deliver your study medication.

Your infusions will be given using an infusion pump and an inline filter. An infusion pump is a device that delivers medications into your body at a controlled rate. An inline filter is a small filter in the plastic tubing used to prevent bacteria and other unnecessary or unwanted materials from getting into your body. Each IV infusion of study medication will take about <u>2 hours</u>. If you have side effects that appear to be related to how quickly the study medication is being infused, it may be given to you more slowly, about 30 minutes or 1 to  $1\frac{1}{2}$  hours longer, depending on what your study doctor thinks is most safe.

#### How often will the study medication be given to me?

Study medication will be given once every 3 weeks. This means that study medication will be given on Day 1 of each 21-day period. Each of these 21-day (or 3 week) periods is referred to as one "cycle" of dosing.

# Will I need to stay in the hospital during this study?

No, it is not expected that you will need to stay in the hospital during this study. Administration of study medication, and all the tests and procedures associated with this study can be done on an outpatient basis, meaning you will need to come to the clinic to be seen by the study doctors and study team, but you will not need to stay overnight, unless you have a side effect and the study doctors think staying in the hospital will be safer for you.

#### How will the study doctor know if I have side effects?

The first time you are given the study medication (on Cycle 1/Day1), you will be observed for a minimum of 2 hours after the end of infusion. For all later doses (Cycle 2 and beyond) you will be observed for a minimum of 1 hour following the infusion.

During Cycle 1, which will be the first 3 weeks you are on study, and throughout your participation in this trial, your doctor will ask questions about how you are feeling and whether you are having any side effects. In addition, throughout the study your doctor will carefully monitor your condition by physical exams, lab tests to check your blood and urine, as well as ECGs to check your heart, pulmonary function tests (also called PFTs) to check your lungs, imaging studies such as chest X-rays to check your lungs, as well as CT scans or MRI scans to further check your lungs and to check the overall status of your disease.

#### Will I receive any medications to prevent side effects?

Yes, you will. Beginning with your first dose of study drug, you will receive standard medications <u>before</u> each dose to reduce the risk of a side effect called an "infusion reaction." You will be given these medications also referred to as "premedication", to take by mouth before each infusion. You will need to take a dose by mouth about 12 hours and another dose about 6 hours before your scheduled infusion of study drug. In addition, when you arrive at the study center the morning of your infusion, you will be given premedications by IV and perhaps also by mouth beginning at least <u>30 minutes</u> before each infusion of study drug. There are more details about infusion reactions later in this consent form.

## What will happen if I have other side effects?

At the first sign of unacceptable side effects, your doctor may decide to prescribe additional medications to treat or attempt to prevent the side effects.

In addition, study medication dosing may be interrupted (stopped temporarily), dosing may be slowed (your 2 hour infusion may be stretched to a longer period), the dose may be lowered, or the dosing may be stopped completely at any time if you experience any side effects during the treatment periods that suggest such actions may help you. If necessary, your doctor may decide to remove you from the study.

# How many cycles of study medication will I receive?

At the end of the first cycle, if you are experiencing no significant side effects, you will go on to receive an additional cycle. Your doctor will monitor your condition carefully throughout this period.

As the study progresses, the number of cycles you will receive will also depend on the results of imaging studies (scans) performed to assess the status of your disease.

• At the end of 2 cycles (after receiving 2 doses [after 6 weeks]), and every 2 cycles (6 weeks) thereafter, you will have imaging studies performed.

At these points, if you agree, and if there is evidence that the study treatment may be improving or stabilizing your disease, your doctor may recommend that you continue to receive additional cycles. You may continue receiving cycles of study medication as long as your doctor recommends, as long as you consent to participate, and as long as your disease is not progressing and requiring alternative therapy, provided you are tolerating any side effects from the study medication.

#### How many hospitals and how many patients will take part in this study?

It is expected that about 90 patients in total will participate in this study.

- Part 1: The initial part of this study took place at 2 different clinics in the United States (U.S.). 24 patients participated in this part of the study.
- Part 2: This part of the study will take place at approximately 6 to 12 clinics in the U.S. and Canada. Approximately 60 patients will participate in this part of the study.

#### 3. TAKING PART IN THE STUDY

It is up to you to decide whether or not to take part in the study. You are free to refuse to participate. Even if you refuse to participate in this study, you will not be disadvantaged in any way. Your refusal will not affect the medical treatment and care you are entitled to receive. If you decide to participate, you may change your mind and decide to withdraw from the study at any time and for any reason. You are not required to explain your reasons for withdrawing. If you withdraw, you will not suffer any penalty or loss of benefits regarding your future care.

Your study doctor can also withdraw you from the study at any time if he or she feels it is in your best interest, or if you cannot comply with study requirements.

In addition, your participation in the study may be stopped by the Sponsor, by regulatory authorities, or by your hospital's independent Institutional Review Board (IRB) or independent research Ethics

Committee (EC) (The IRB or EC is responsible for reviewing the design and approving the ethical conduct of this study in order to assure that patient safety is maintained and patients' rights are not violated) at any time without your consent. If this were to happen, it would occur after the reason(s) for doing so has been explained to you, and after you have been given advice about continued care for your condition, if this is appropriate.

Also, the Sponsor has the right to stop the study for medical or business reasons. If this happens, all patients participating in the study will be withdrawn.

If you withdraw (or are withdrawn) from the study, you will be asked to go through End of Treatment and One Month Follow-up procedures detailed later in this consent form.

#### 4. STUDY PROCEDURES

## What tests and procedures will I undergo as part of this study?

If you agree to participate in this study, first you will have several tests and procedures done to see if you qualify for the study, and if it is safe for you to participate. This is called the "Screening" process. During Screening for this study, your doctor will ask you many detailed questions about your medical history, about your disease and other treatments you may have received for it, and about other medications you have taken or are now taking.

During Screening, as well as throughout the study, your doctor will carefully monitor your condition by asking you questions about how you are feeling. You will also have the following tests and procedures performed at Screening and at different times during the study (times that will be detailed later in this consent form):

- Your doctor will measure your height, weight, check your vital signs (temperature, blood pressure, heart rate, and oxygen content in your blood), perform physical exams always including an assessment of your lungs, an eye exam, and lab tests to check your blood and urine.
- If you are a woman who is capable of getting pregnant, you will have pregnancy tests done. These tests must be done on a blood sample at screening, but may be done on a blood or urine sample when repeated later in the study. If you are a woman capable of getting pregnant, or a man in a relationship with a woman capable of getting pregnant, the doctors will explain to you how important it is for a pregnancy not to occur during the study and for a period of at least 3 months after you have taken your last dose of study medication. The doctors will then counsel you on how best to avoid pregnancy during this period.
- The condition of your heart will be checked by measuring the electrical traces of your heart, a painless procedure called an electrocardiogram (ECG). In addition, you may have another heart test, either an echocardiogram ("Echo") or a multigated acquisition (MUGA) scan, to further check the condition of your heart and to assess how well your heart is working as a pump. These tests will be described in more detail later in this consent form.
- The condition of your lungs and how well they are working will be checked by pulmonary function tests (PFTs). These tests will be described in more detail later in this consent form. You will also have chest X-rays to check the status of your lungs.
- Your study doctor will perform tests to check the status of your disease. You will have imaging tests (such as a CT scan or MRI scan) to check the location and size of your cancer. Whatever

test your doctors use to check your disease at the beginning of the study will most likely be the same test that will be used later during the study. The choice of test will depend on your disease type because different tests are better for checking different diseases. These tests will also be used to check the status of your lungs.

- Your doctor will ask to evaluate a left-over sample of your tumor that has been stored (archived) after a previous biopsy or surgery to determine whether your tumor cells are positive for the target of this study medication. In addition, other tests called "biomarker tests" will be done to learn more about the tumor. Your study doctor will talk to you about arranging to get a small portion of that sample sent in so these tests can be done.
  - Tumor testing is <u>required</u> because **your tumor must be positive for the target of this study medication** in order for you to participate. Tumor samples will be sent to a central lab for this testing.

If a sample of your tumor is not available, or if there is not enough tumor tissue to do all the required testing, you will be asked to have a biopsy of your tumor performed. If this is the case, you must be willing to undergo this biopsy in order to determine whether you will be eligible to participate in the study. If such a biopsy is necessary, the study doctor will discuss this with you.

A tumor biopsy is a procedure in which a small sample of your tumor is removed with a thin needle. You will be asked to agree to this procedure only if your doctor thinks your tumor is safely accessible for biopsy and it is thought that such procedure can be done with minimal risk to you. You will receive a painkiller prior to the biopsy and/or some anaesthesia to numb the area where the needle will pass. This procedure will be described in more detail later in this consent form.

The following tests and procedures will also be performed during the study, but <u>only</u> after it is determined that you qualify for the study and it is considered safe for you to participate:

- You will undergo blood tests that will help the doctors determine how the study medication is
  absorbed by your body and how long it stays in your blood. These are called "pharmacokinetic
  studies", or "PK studies." Blood samples will be sent to a central lab for this testing. If there is
  blood left over from these tests, the blood may be used to do some of the "biomarker tests"
  mentioned above.
- You will have blood tests to check whether your body has made antibodies (proteins made by the immune system) to the study medication. These are referred to as "anti-drug-antibody (ADA) tests." Blood samples will be sent to a central lab for this testing. Once again, if there is blood left over from these tests, the blood may be used to do some of the "biomarker tests" mentioned above.
- Your study doctor will ask for a blood sample to do "biomarker tests" on tumor cells that may be circulating in your blood. If you have a cancer of the **head or neck**, additional tests will be done on this sample.

# Will all patients participating in the study undergo the same tests and procedures?

All of the tests listed are required, meaning if you participate in this study you must agree to have all of them performed.

#### Are there other tests that may be performed that are not required, but are considered optional?

Yes, there is optional testing that may be requested of you. This testing involves collection of tumor tissue for "biomarker tests." You may refused these tests and still be eligible to participate in this study. The conditions for this optional testing are as follows:

- Should you require surgery on an area of tumor while you are on this study, the doctors will ask your permission to submit a small portion of the tumor tissue for testing.
- Should you have a response to the study medication while you are on this study, or should you have a period of no growth of your tumor for more than 8 weeks, the doctors will ask your permission to biopsy an area of tumor that remains in order to submit the tumor tissue for testing.
- Should other study findings suggest that more could be learned about the study medication if your tumor could be tested after dosing, the doctors will ask your permission to biopsy an area of tumor in order to submit the tumor tissue for testing.

#### How much blood will be taken from me during this study?

Routine blood tests require a little more than 1 tablespoon of blood. One tablespoon of blood is equal to about 15 milliliters (mL), and routine blood tests require about 20 mL, although efforts will be made to collect smaller amounts of blood for these studies where possible.

In addition, each PK test requires a teaspoon (5 mL), and a pregnancy test (if you should need one), and the anti-drug antibody test each require about 1 teaspoon each (about 5 mL).

Throughout the study, blood will be taken on all study visit days, but the most blood that will be taken from you on any day will be as follows:

- <u>Screening</u>: a little less than 2 tablespoons (about 25 mL)
- Cvcle 1
  - o <u>Day1</u>: When PK samples will be taken, a little more than 2 tablespoons (about 35 mL)\*
  - O Day 4: A little more than 1 tablespoon (about 20 mL)
  - O Day 8: A little less than 2 tablespoon (about 25 mL)
- Cycles that Follow
  - O Day 1: About 3 tablespoons (about 45 mL)
  - o <u>Day 8</u>: A little more than 1 tablespoon (about 20mL)
- Cycles that Follow except Cycle 5
  - o <u>Day 1</u>: A little more than 3 tablespoons (about 50 mL)
  - o <u>Day 8</u>: A little less than 2 tablespoons (about 25 mL)
- End of treatment visit: about 2 tablespoons (about 30 mL)\*
- One month follow-up visit: about 2 tablespoons (about 30 mL)

• In addition, if you should have an infusion reaction a little more than a teaspoon of blood will be taken (about 10 mL for PK and ADA studies) to be tested so that more can be learned about the study medication during these reactions.

\*Patients with cancer of the **head or neck** will have a little more than 1 tablespoon extra taken on these days
The total amount of blood taken from you will depend upon how long you remain on the study; cycles after Cycle 1 require a little less blood to be taken.

#### 5. SCHEDULE OF TESTING DURING THE STUDY

You must agree to come to the study center on the days specified by your study doctor, so that the necessary tests can be done. Your study doctor and his or her staff will give you a schedule that lets you know when you need to come to the center and will explain what tests will be performed at each visit. Most of the tests that will be done throughout the study are routine tests that are part of the normal care of patients with your condition. What you can expect at each point of the study is described below.

## **SCREENING**

If you decide to participate, and after you sign this informed consent form, the following tests and procedures will be done to make sure it is safe for you to take part in the study. Most of these tests will be done within 14 days before you receive the first dose of study medication, some may be done within 28 days before you receive the first dose. The screening process may take more than one day to complete.

- Review of your past medical history: You will be asked several basic questions (for example, your gender, age, and ethnicity). You will be asked about your past and current health problems and about any prior surgical procedures you have had that are not related to your disease.
- Review of your cancer history: You will be asked about the prior surgical procedures you have had that are related to your disease and about the cancer therapies you have received for your disease.
- Review of your current medications: You will be asked about the medications you use currently as of the day of screening, including vitamins, nutritional supplements, or herbal medications not prescribed by your doctor.
- Performance status: You will be asked to rate how well you can carry out your normal daily activities (this is called performance status).
- Vital signs: You will have your temperature and vital signs (including your pulse, breathing rate, blood pressure, and oxygen concentration in your blood) measured to check your overall health.
- Physical exam: You will have a complete physical examination including an assessment of your general appearance and measurement of your height and weight.
- Eye exam: You will have an exam of your eyes, including an evaluation of your corneas, which are the transparent layers that form the front of the eyes.
- Routine blood and urine tests: Blood and urine will be collected for routine laboratory tests.
- Pregnancy test: If you are a woman who may be able to get pregnant, a pregnancy test will be done. The results of this test must show that you are not pregnant in order for you to take part in

this study. This test must be done on a blood sample at screening, but may be done on a blood or urine sample when repeated later in the study

- ECG: You will have an electrocardiogram done; this is an electrical tracing of your heartbeat.
- Echo or MUGA: Either you will have an Echo or a MUGA scan to check the activity and function of your heart, but only if you have a history of heart problems.
- Pulmonary function tests: You will have a group of tests that measure how well your lungs work.
   This includes how well you are able to breathe, and how well your lungs are able to bring oxygen to the rest of your body.
- Chest X-ray: A chest x-ray will be done to check the condition of your lungs.
- CT scan or MRI: You will have either a CT scan or an MRI to check the status of your disease (unless you have had one of these scans within 28 days of the screening visit and the results are made available to the study doctor).
- Stored (archival) tumor sample or tumor biopsy: A request will be made to obtain a sample of your tumor tissue from a previous biopsy or surgery to determine whether your tumor is positive for the target of this study medication and to do biomarker studies.
  - O Providing a sample of tumor tissue is required, and if not available, you will need to undergo a biopsy to collect tumor tissue for testing. The test performed must show that your tumor is positive for the target of this study medication for you to be eligible for the study, and there must be enough tumor tissue to perform the other required biomarker studies.

Once it is confirmed that you are eligible for the study, and it is safe for you to take part, the following will be done:

• A blood sample will be taken to do tests on tumor cells that may be circulating in your blood

#### STUDY MEDICATION SCHEDULE

If your Screening tests show that you can take part in this study, you will receive the study medication into your vein (IV) on Day 1 of each 21-day (3-week) cycle. Your study doctor will also provide you with premedications to take by mouth. You will take these medications at home about 12 hours and about 6 hours before each of your scheduled infusions of study drug.

# STUDY VISIT SCHEDULE

#### Cycle 1

<u>Day 1</u>: On the first day of dosing, you will need to remain at the clinic, until about 2 hours after your study medication infusion is completed.

Several blood samples will be taken on this day, so a member of the study team will insert a catheter (a thin, flexible tube also called "an IV") into one of the veins (probably in your arm) so you won't need to be stuck with a needle many times to take the samples.

During this visit <u>premedication will be administered</u> and the following will be done:

Items that are italicized: may not need to be repeated if you had your Screening visit within 7 days before starting the study medication

- Review of your medications and review of any symptoms that you may be experiencing or have been experiencing since the last visit
- Vital signs
- Physical exam including body weight and lung assessment, and assessment of your performance status
- Routine blood and urine sample collections to check your overall health
- Pregnancy test if you are a woman who may be able to get pregnant required within 2 working days of receiving your first dose
- PK blood sample collection one sample before getting your study medication dose, and one at the end of infusion
- ADA blood sample collection to compare to samples that will be taken later in the study to check whether your body has made antibodies to the study medication
- Premedication administration
- Study medication administration

#### Day 4: During this visit the following will be done:

- Review of your medications and review of any symptoms or side effects that you may be experiencing or have experienced since the last visit
- Routine blood and urine sample collections to check your overall health

#### <u>Day 8</u>: During this visit the following will be done:

- Review of your medications and review of any symptoms or side effects that you may be experiencing or have experienced since the last visit
- Routine blood and urine sample collections to check your overall health
- PK blood sample collection one sample

#### Subsequent Cycles

If you tolerated the first cycle and remain on the study, you will continue to receive the study medication on Day 1 of each 21-day (3 week) cycle. During each cycle, you will also need to have the following tests and procedures.

<u>Day 1</u>: During this visit <u>premedication will be administered</u> and the following will be done:

- Review of your medications and review of any symptoms or side effects that you may be experiencing or have experienced since the last visit
- Vital signs
- Physical exam including body weight and lung assessment, and assessment of your performance status
- Routine blood and urine sample collections to check your overall health

- PK blood sample collection one sample before getting your study medication; one sample at the end of infusion during Cycle 5 only
- ADA blood sample collection
- Premedication administration
- Study medication administration

#### <u>Day 8</u>: During this visit the following will be done:

- Review of your medications and review of any symptoms or side effects that you may be experiencing or have experienced since the last visit
- Routine blood and urine sample collections to check your overall health
- PK blood sample collection one sample during Cycle 5 only

## End of Even-Numbered Cycles (Cycle 2, 4, 6, etc.)

<u>During the week prior to Day 1 of the next cycle</u>: During this visit, the following will be done:

- Review of your medications and review of any symptoms or side effects that you may be experiencing or have experienced since the last visit
- CT scan or MRI to assess your disease and check your lung status
- End of Cycle 2 only: Ophthalmology Exam

#### End of Treatment Visit

You will need to return to the clinic within 10 days following the decision for you to discontinue participation in the study to have the following done:

- Review of your medications and review of any symptoms or side effects that you may be experiencing or have experienced since the last visit
- Vital signs
- Physical exam including body weight and lung assessment, and assessment of your performance status
- Eye exam
- Routine blood and urine sample collections to check your overall health
- ADA blood sample collection
- Pregnancy test if you are a woman who may be able to get pregnant
- ECG to check your heart
- ECHO or MUGA to check your heart (only if you have a history of heart problems)
- Pulmonary function tests to check your lungs
- Chest X-ray to check your lungs
- CT scan or MRI to assess your disease and check your lung status (only if it has been more than 6 weeks since the previous CT or MRI)
- PK blood sample collection one sample during visit

• Patients with a cancer of the head or neck: a blood sample will be taken to do tests on tumor cells that may be circulating in your blood

#### One Month Follow-Up Visit

You will need to return to the clinic about 1 month (30 days) after your last dose of study medication to have the following done:

Note: Depending on scheduling and when the decision is made for you to leave the study, the End of Treatment Visit and the One Month Follow-up Visit may be done on the same day. If this is the case, the assessments listed to be performed at the End of Treatment Visit will be the assessments to be conducted.

- Review of your medications and review of any symptoms or side effects that you may be experiencing or have been experiencing since the last visit
- Vital signs
- Physical exam including body weight and lung assessment, and assessment of your performance status
- Routine blood and urine sample collections to check your overall health
- ADA blood sample collection
- CT scan or MRI to assess your disease and check your lung status (only if disease progression was not shown on a previous CT or MRI)
- PK blood sample collection one sample during visit

## 6. POSSIBLE RISKS OF PARTICIPATING IN THIS STUDY

As with all research studies, the study medication and study procedures may involve unknown risks. Any medication can have temporary and/or permanent side effects and can cause unforeseen adverse reactions.

#### What are the risks associated with AVID100?

Little is known about potential side effects of AVID100 since this is the first study in which it is being tested in humans. Based on animal studies conducted in which monkeys were given AVID100, as well as side effects known to occur with drugs similar to AVID100, including antibodies linked to cancer chemotherapy agents, the following side effects have been observed suggesting that some of these effects may be seen in patients treated with AVID100:

#### Side effects of AVID100 in animal studies and of side effects of drugs similar to AVID100:

- Skin changes including:
  - o Generalized rash, acne-type rash, or red/bumpy rash
  - Skin thickening, redness, increased pigment
  - o Dryness, flaking, and/or cracking
  - o Itching and eczema
  - Skin and nail infections
  - Sores, scabs, bruises, ulcers, changes in healing
- Fatigue, weakness
- Headache
- Diarrhea, constipation, abdominal pain

- Dehydration
- Loss of appetite, weight loss
- Rapid heartbeat, slowed heartbeat, irregular heartbeat
- Unusual taste in the mouth
- Swelling of the face
- Inflamed lips and membranes of the mouth causing sores and pain
- Inflamed membranes of the eye causing redness and pain
- Blistering and swelling of the hands and feet
- Changes in blood tests, particularly:
  - O Decreases in red blood cells which could cause anemia, the symptoms of which are tiredness/fatigue, and shortness of breath
  - Decreases in platelets (which help the body with blood clotting), which could result in increased bruising and longer bleeding from a cut or injury, including excessive bleeding (hemorrhage)
  - o Decreases in blood salts (called electrolytes) such as magnesium, calcium, and potassium
  - o Increases in tests that measure how the liver is working
- Damage to the nervous system resulting in numbness, tingling, and weakness in the arms, hands, legs, and feet (also known as peripheral neuropathy)
- Damage to the liver, including liver failure
- Damage to the lungs, including scaring and stiffness of the lungs (a condition called pulmonary fibrosis)
- Abnormalities in tissues when looked at under a microscope, including changes to the:
  - Eyes, particularly the layers that cover the front of the eye (the cornea and the conjunctiva), which could mean the eyes are being damaged
  - o Bone marrow, where there could be a decrease in cells that make the blood
  - o Thymus and lymph nodes, where there could be fewer cells to help the immune system
  - Ovaries (in women), which could result in changes in fertility
  - o Sperm (in man) where there could be a decrease in number
  - o Skin, liver, heart, GI tract changes suggesting inflammation and damage

#### What other risks can be anticipated with AVID100?

Along with the side effects listed above, because you will be receiving the study medication by intravenous (IV) infusion, there is a risk of experiencing what is called an **infusion reaction**.

Infusion reactions have been seen with other drugs that are similar to AVID100, and even though the risk of these reactions does not appear to be as great with AVID100, having such side effects is still possible. You will be given medications to try to decrease or prevent these reactions before receiving an AVID100 dose. Infusion reactions may include:

#### Side effects of infusion reactions:

- Facial flushing and/or swelling
- Rash
- Fever
- Shortness of breath
- Wheezing
- Headache
- Nausea
- Dizziness
- Sweating
- Feeling anxious
- Fast heart rate
- Low blood pressure
- Chills and/or cold sweats
- Chest and throat tightness
- Airway spasm
- Chest, back, and/or abdominal discomfort/pain

#### What is the experience thus far with AVID100 in this study?

Thus far, a limited number of patients have been treated with AVID100 in this study, so a limited amount of information is available. The side effects that have been seen thus far are listed below.

## Side effects of AVID100 seen in this study (mostly mild to moderate in severity)

Side effects seen most often have included (in 20% or more of patients):

- Rash and acne-like rash
- Fatigue
- Nausea
- Decrease in platelets (which help the body with blood clotting), which could result in increased bruising and longer bleeding from a cut or injury, including excessive bleeding (hemorrhage)

#### Side effects seen less frequently have included (in 5% to up to 20% of patients):

- Infusion reactions
- Headache
- Vomiting
- Diarrhea
- Not feeling hungry
- Mouth sores
- Dry skin
- Itching
- Redness/itchiness of the eyes
- Irritation of the cornea, which is the transparent layer forming the front of the eye
- Watery eyes
- Cough
- Decrease in red blood cells which carry oxygen to tissues and may result in tiredness and shortness of breath
- Increase in blood chemicals that are measures of how your liver is doing
- Increase in blood lipase, a chemical involved in digestion and a measure of how your pancreas is doing
- Decreases in electrolytes, which are the salts in the blood
- Protein in the urine which could be due to kidney injury

## Side effects seen rarely have included (in less than 5% of patients):

- Dry eyes
- Eye pain
- Eyes sensitive to light
- Inflammation of the cornea and deeper layers of the eyes
- Bloody nose

# Side effects of AVID100 seen in this study (mostly mild to moderate in severity)

- Increased sweating
- Feeling of discomfort
- Abdominal pain
- Dehydration
- Altered sense of taste
- Weight loss
- Hair loss
- Muscle aches
- Restless legs
- Numbness and tingling in the hands and feet
- Lung inflammation
- Shortness of breath
- Decreased amount of air breathed out during breathing tests
- Worsening asthma symptoms
- Irritation of the sinuses
- Cold-like symptoms
- Flu-like symptoms
- Poor wound healing
- Infection of the mouth
- Dry mouth
- Fungal infection of the skin
- Bladder infection
- Decrease in white blood cells called lymphocyte which help the body fight infection
- Change in a blood test that measures how long it takes blood to clot
- Increase in blood amylase, a chemical involved in digestion and a measure of how your pancreas is doing
- Increase in blood uric acid, a measure of how your kidney is doing
- Decrease in blood albumin, a protein made in the liver that helps keep body fluids in balance

#### More severe side effects have been rare and have included (in less than 5% of patients):

- Vomiting (at a dose higher than is being given in the Phase 2 part of this study)
- Decrease in lymphocytes with no symptoms
- Decrease in platelets with no symptoms
- Increase in blood chemicals of liver function with no symptoms
- Increase in blood lipase with no symptoms
- Protein in the urine with no symptoms
- One patient experienced sores in the mouth that were considered severe. When healed the patient continued on study at a lower dose.
- Two patients experienced pneumonitis, which is an inflammation of the lungs. It was considered severe in both cases. In one patient it was accompanied by shortness of breath, cough, wheezing, painful breathing, and decreased oxygen levels in the blood. The patient was taken off study, treated with steroids, and was reported to improve. In the second patient it was accompanied by shortness of breath, anxiety, extreme fatigue, and decreased oxygen levels in the blood. Symptoms began after the patient was off study and were reported to be resolving.
- One patient experienced a decrease in platelets, which help the body with blood clotting. The patient then had a fall
  hitting his head which resulted in bleeding in his head. The patient recovered and continued on study at a lower
  dose.
- One patient experienced an infusion reaction that was considered severe, with shortness of breath, chest tightness, chest pain, and rapid heartbeat reported. The infusion was stopped; the patient was given medications and watched carefully at the clinic and briefly at the ER until the symptoms went away. The patient was taken off the study. This patient received study drug by a shorter infusion time (1 hour) than is used now (2 hours); and was treated at a point in the study when premedications were not required to be given
- One patient experienced an infusion reaction that was considered life-threatening, with shortness of breath, and
  difficulty breathing. The infusion was stopped; the patient was given medications, taken to the hospital, and
  required a breathing tube. The patient was taken off the study and recovered from the reaction.

#### Side effects of AVID100 seen in this study (mostly mild to moderate in severity)

If you should have an infusion reaction, 2 blood samples will be taken (about 1½ teaspoons) so that PK and ADA tests can be done in an effort to better understand these reactions.

# What will be done to prevent or lessen side effects from the study medication and what should I do if I have side effects?

All care will be taken to minimize side effects, but they can be unpredictable both in nature and severity. In order to ensure that your treatment is as safe as possible, you will be watched carefully throughout each infusion of study medication, and for a period of time following each infusion until it is considered safe for you to leave the clinic. After your first infusion, you will be monitored for at least 2 hours after the end of your infusion. For each subsequent infusion, you will be monitored for at least 1 hour after the end of your infusion. Throughout the study, your doctor will ask questions about how you are feeling and whether you are having any side effects. In addition, your study doctor will carefully monitor your condition by physical exams, frequent blood tests will be done, and special attention will be paid to the workings of your eyes, heart, lungs, kidneys, liver, and digestive system.

Medicines or supplements you might be taking could cause side effects if you use them while you are receiving AVID100. Because of this, you must tell your study doctor or a member of the study staff about all your past and present illnesses and allergies. You must also tell them about all vitamins, supplements, and medicines you are taking.

For your own safety and for the safety of other participants in the study, you must inform the study doctor or study staff about any side effects or other health problems you experience during the study. This should be done, no matter how minor the changes might seem to you, whether or not you think they might be caused by the study medication.

Any side effects that may occur during treatment need to be carefully monitored by your study doctors so that they can give you the care that you need. You will be given premedications before your dose(s) of study medication to decrease or prevent these side effects; however, if the doctors see a pattern in any other side effects that you experience during this study, they may give you additional medications before you receive your dose(s) in an effort to lessen the side effects or prevent them from occurring.

At the first sign of any unacceptable side effect, you will be given medication to treat your symptoms. In addition, your doctor may decide to interrupt, slow, lower, or stop your dose, or it may be necessary to remove you from the study. If stopped and restarted, your infusion may be given to you at a slower rate.

#### What are the risks associated with pregnancy during this study?

If you become pregnant, or if your partner becomes pregnant, there may be unknown risks to the embryo or fetus. If you are a woman who is able to have children (unless you have had a hysterectomy, tubal ligation, or you have been postmenopausal for at least one year) you will have a pregnancy test at screening, and if the result is positive, you will not be able to be in the study.

If you are a sexually-active man or woman, you must use a medically effective form of birth control as per institutional standards throughout the study and for <u>3 months</u> after the last dose of study medication. The study doctor will discuss methods of birth control with you, if needed.

If you become pregnant or think you may be pregnant during the study, contact the study doctor's office **immediately**. You will be withdrawn from the study. If your partner becomes pregnant or thinks she may be pregnant during the study, contact the study doctor's office **immediately**.

The study doctor must follow up and document the course and the outcome of all pregnancies, even if you withdraw from the study or if the study has finished. If you or your partner becomes pregnant during the study, the study doctor or his/her staff will ask to contact you/your partner and your/your partner's physician for information about the pregnancy and the child until at least 3 months after the birth. You must not be breast-feeding during the study.

#### Are there other risks associated with taking part in this trial?

A possible concern is that there may be a risk associated with <u>other medications</u> you might be taking while on this trial. Since there is no way to predict whether the study medication might interact in some way with other drugs or medications, it is very important that you tell your study doctor all the medications you take throughout the entire time you are on the study. Your study doctor will ask you questions about this at each visit.

In particular, there is a concern about taking <u>herbal medications or preparations for your cancer</u>, such as those that are available at health food stores to treat disease and improve well-being. These medications and preparations <u>should not</u> be taken while you are on this study because there is no way to determine how they will affect you or the way the study medication is handled by your body.

#### What are the risks associated with study procedures?

<u>Blood sampling</u>: Blood will be taken from a vein in your arm during the study. The taking of a blood sample may cause some discomfort and bruising, and there is a potential for infection. Other risks, although rare, include dizziness and fainting.

<u>IV catheter placement</u>: On days of multiple PK sampling, an IV catheter may be placed in order to reduce the number of times you would need to be stuck with a needle. If you have a catheter or port in place, consideration may be given to using this for IV access to deliver the study medication.

<u>Blood pressure</u>: An inflatable cuff will be placed on your arm, and a machine will measure your blood pressure and heart rate. You may experience mild discomfort in your arm while the cuff is inflated.

<u>Electrocardiogram (ECG)</u>: This is a painless, non-invasive test that shows how your heart is working by making a tracing of the electrical activity of your heart. To have an ECG, you will lie on a bed/couch for several minutes. Small sticky pads called electrodes will be stuck to your chest, shoulders and hips (or ankles) and a machine will measure the electrical activity of your heart. Small patches of your hair may need to be clipped in these areas. The sticky pads may cause some local irritation and may be uncomfortable to remove.

Echocardiogram (ECHO) (only in patients with a history of certain heart problems): An Echo is an ultrasound of your heart. Gel will be spread on your chest and then a device known as a transducer will be pressed firmly against your skin, aiming an ultrasound beam through your chest to your heart. The transducer records the sound wave echoes from your heart. A computer converts the echoes into moving images on a monitor. You may feel uncomfortable from lying still or from the transducer pressing on your chest.

Multigated acquisition (MUGA) scan (only in patients with a history of certain heart problems): A MUGA scan creates video images of the heart to see how it is working. A special camera will be used to monitor your heart's activity during the test. Electrodes will be placed on your chest to monitor your heart's electrical activity during the test. A small amount of radioactive material, called a tracer, will be injected into a vein in your arm. Sometimes a small amount of blood from your arm will be withdrawn and mixed with the tracer. Then the mixture will be put back into your body through the vein. Similar to taking a blood sample, there may be some discomfort and bruising where the needle was inserted, and there is a potential for infection. Other risks, although rare, include dizziness and fainting. There is also a slight risk of allergic reaction to the radioactive tracer.

<u>Pulmonary function tests (PFTs)</u>: These tests determine how much air your lungs can hold, how quickly you can move air in and out of your lungs, and how well your lungs put oxygen into and remove carbon dioxide from your blood. You will need to breathe into a mouthpiece attached to a recording device (spirometer). You will also need to take a breath of air containing a very small amount of carbon monoxide while measurements are taken from the breath you exhale. There should be no pain or discomfort involved in these tests.

Computerized tomography (CT) scan: A CT scan is a series of cross-sectional X-rays of your body. CT scans do expose you to more radiation than a standard X-ray, but the risk is small. Some people have a reaction to the contrast dye that is injected into a vein before the scan, as it contains iodine, so you will have to tell your doctor if such a reaction has ever happened to you in the past. Allergy to iodine may cause nausea, vomiting, sneezing, itching or hives. A severe allergic reaction (called anaphylaxis) that results in difficulty breathing can occur, but it is rare.

Magnetic resonance imaging (MRI): An MRI scan is painless and will not expose you to X-ray radiation. Before this scan, contrast medium may be injected into one of your veins; this is like a dye and will spread through your body and will help give clearer images. The injection of contrast medium may cause some discomfort and bruising. There is a risk of potentially serious reactions in some individuals who receive contrast medium. Some people may feel frightened by the cramped space inside the machine or by the loud, repeated sounds the machine makes. The greatest risk of having an MRI is the chance of metal objects moving rapidly toward the magnet and hitting you. To reduce this risk, all people giving and getting the MRI scan will be asked to remove all metal from their clothing and all metal objects from their pockets. Please inform the study doctor if you have metal in your body from an operation, since you may not be able to have a MRI scan. Also, if you have a pacemaker you should not have a MRI scan.

<u>Tumor biopsy</u>: A tumor biopsy is a procedure in which a small sample of your tumor is removed with a thin needle. You may be asked to agree to this if samples of your tumor are not available from a previous biopsy or surgical procedure, but only if the study doctor thinks your tumor is safely accessible for biopsy. A tumor biopsy is done to diagnose and gather information on a tumor or potential tumor. You will receive a pain-killer prior to the biopsy and/or some local anesthesia to numb the area where the needle will pass to help control any discomfort or pain. You may also be given medications to make you sleep during the procedure.

There are general risks that are part of any surgery procedure, no matter how minor, such as: excessive bleeding; infection; damage to nearby organs; discomfort or pain at the biopsy site; delayed healing at the biopsy site; reactions from pain medications which may include constipation, sluggishness and fatigue, or dry mouth; reactions from anesthesia which may include drowsiness, dizziness, confusion, shakiness,

ringing in the ears, nausea, tingling or numbness, visual changes, slurred speech, muscle twitching, changes in heartbeat, decreased blood pressure, and extremely rarely seizures or severe and dangerous blood pressure changes; more serious reactions, may occur rarely.

#### 7. POSSIBLE BENEFITS OF PARTICIPATING IN THIS STUDY

You may not get any direct benefit from taking part in this study. You will be given close attention from the study staff during the time you are involved in the study. You may receive information about your health from physical examinations and medical tests done in this study.

This study is expected to benefit the Sponsor by providing information on whether the study medication might be a useful treatment for patients with certain epithelial solid tumor cancers.

If the results of this study are favorable, and, along with additional studies that lead to approval by regulatory authorities of AVID100 for use in humans, there may be benefits for patients in the future.

#### 8. ALTERNATIVE TREATMENTS

You do not have to be in this study to get treatment for your cancer. Instead of taking part in this study, your doctor will explain the other options available to you. These options may include:

- Receiving other treatments for your cancer, if such treatments are available.
- Taking part in another research study
- Getting no treatment for your cancer, or
- Receiving "comfort care only" where treatments are directed only at reducing symptoms, relieving suffering and maximizing comfort, dignity, and control. In comfort care only, treatment is not directed at curing, slowing, or reversing your disease.

If you have any questions concerning alternative treatments, please ask your study doctor. Your study doctor can discuss your treatment options with you. If you decide not to take part in this study, your decision will not affect your care at this hospital.

#### 9. COSTS RELATED TO THE STUDY

Study medication will be provided at no cost to you. In addition, there will be no cost to you for the additional blood and urine tests, hospital stays, doctor visits, and other procedures related to this study.

You, your insurance company, or government program, are responsible for the costs of the usual tests and procedures done in the routine care for your cancer. This includes the cost of routine blood and urine tests, x-rays, scans, surgeries, other treatments, and physician's charges that are not related to this study.

#### 10. COMPENSATION RELATED TO THE STUDY

You will not receive any financial compensation for taking part in this study.

This study is part of the development of a potential new drug. If the results of the study are successful, and the study medication is eventually sold commercially, you will not be compensated for taking part in this study.

AVID100-01: Model ICF: Version 5.0 30May2020 (P2 stand-alone)

#### 11. INJURY OR COMPLICATIONS

If you suspect illness or injury you should contact your study doctor immediately. In the event of illness or injury resulting from your participation in this trial, necessary medical treatment will be provided.

If not covered by your insurance, government program, or by any other third party, the Sponsor will pay for such emergency medical treatment and will provide payment for reasonable medical expenses, including hospitalization, subject to the treatment being required as a direct result of the study medication or its administration in accordance with the Protocol, as determined by the Sponsor and the study doctor. No other type of compensation such as lost wages or other damages will be paid to you as a result of your taking part in this study.

The Sponsor will not provide payment for expenses that are in any way attributable to the negligence or misconduct of any person employed by or acting on behalf of the Investigator or the Site. The Sponsor will not pay for medical expenses for injuries unrelated to the study medication or which are in any way attributable to known or expected side effects or to the natural course of any underlying disease or treatment process.

If you have any questions concerning the availability of medical care or if you think you have experienced a research-related illness, injury or emergency, contact:

| (insert name and telephone number of appropriate contact) |
|-----------------------------------------------------------|
| Contact Name: |
| Telephone Number: |

#### 12. **NEW INFORMATION**

If any new information about the study medication becomes available which may influence your decision to continue in the study, you will be told in a timely manner so that you can decide whether to withdraw from the study.

#### 13. REMOVAL OR WITHDRAWAL FROM THE STUDY

You may be removed from the study without your consent if you experience a side effect or develop a medical condition during the study that your doctor thinks may put you at serious risk. You may be removed from the study without your consent if your doctor decides that your disease has worsened and the treatment is not providing benefit.

You have the right to withdraw from the study at any time. If you are removed or decide to withdraw from the study, you are entitled to receive treatment according to the standard of care for your medical condition as determined by your doctor. Should you be removed from the study, or if you decide to stop taking part in the study, you will be asked to make a final visit to receive physical examinations and to have final laboratory tests performed.

#### 14. TERMINATION OF THE STUDY

In addition to previously mentioned reasons for withdrawal from the study, your participation in this study may be ended without your consent for the following reasons, including:

- If the study doctor believes, for any reason, that it is in your best interest
- If you refuse to have tests that are needed to determine whether this treatment is safe
- If you refuse to have treatment or do not return for follow-up as recommended by your study doctor, or do not follow the study doctor's instructions
- If you require treatment with medications that are not allowed in this study
- If you become pregnant
- If other causes prevent you from continuing in this study
- If the Sponsor decides to end the study or your participation at any time

#### 15. USE OF SAMPLES COLLECTED

The samples that you donate, and related information gathered from the samples, may be provided to the Sponsor and/or its representatives, collaborators, contractors and service providers for analysis in connection with the Study and the development of AVID100. Your samples will not bear your name or any personal information about you, only your study code number will be displayed. During the testing process, any blood or tissue samples collected from you as part of this study will not be used for any other research or genetic tests without your written permission, except for tests specified by the study protocol.

In the future, people who do research with your samples may need to know more about your health. While the doctors coordinating this study may provide reports about your health, they will not provide your name or any other information that will let the researchers know who you are.

The samples collected during this study will be kept until they are used up, or they will be stored for a number of years (possibly up to 15 years) after the end of the study, and will then be destroyed by the laboratory, whichever comes first (the end of the study occurs when a final study report is completed by the Sponsor). The samples will be used for research purposes only and will not be sold.

# 16. CONFIDENTIALITY AND AUTHORIZATION FOR DISCLOSURE

By signing this form, you consent to the study doctor and his or her staff collecting and using your personal data for the study. This includes: your date of birth (day, month and/or year as allowed by local regulations), your sex, your ethnic origin and information on your physical or mental health or condition.

The information shared with the Sponsor is protected by the use of a code, which is a number specifically assigned to you. The study doctor is in control of the code needed to connect your data to you. The Sponsor will not be given your name, but will only know of your code number.

All medical records and research materials that identify you by name will be held confidential (confidential data) so far as permitted by law. However the study doctor, the Sponsor and its representatives, the study monitor (who checks how the study is going and makes sure that the information is being collected properly) and, under certain circumstances, the regulatory authorities and the IRB or EC will be able to inspect confidential data that identify you by name.

All personal data from this study will be treated in accordance with national and local data protection laws.

By signing this consent form, you grant permission for medical information about you obtained during this study (your study data) to be made available to authorized representatives of the regulatory authorities and other government agencies. You also grant permission for your study data to be made available to the Sponsor, the study monitor, other study personnel, and the IRB or EC. The Sponsor may transfer your study data in or outside <u>insert country where study is being conducted</u> for the purposes described in this document. Please be aware that the laws in other countries may not provide the same level of data protection and may not stop your study data from being shared with others. The study doctor, the regulatory authorities, and the Sponsor may keep the study data indefinitely.

You have the right to request information about your study data held by the study doctor and the Sponsor. You also have the right to request that any inaccuracies in such data be corrected. If you wish to make a request, then please contact the study doctor, who can help you contact the Sponsor if necessary.

If you withdraw your consent for participating in this study, your study data that were collected before you withdraw your consent may still be used as described above. Once you have withdrawn your consent for participating in the study, no further data will be collected about you for the purposes of this study unless you agree otherwise, for example, you agree to have further tests and examinations. If you do agree to have further data collected after you have withdrawn your consent, these study data may also be used as described above.

The results of this study may be published in a medical journal and shown at medical meetings. You will not be identified (by name or any other means, e.g., photo) in any of these publications.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law, or in one or more other public trial registries. Such Web sites or registries will not include information that can identify you. At most, they will in include a summary of the trial design and/or a summary of results. You can search these Web sites at any time.

Your health information cannot be used or disclosed (made known) by your study doctor for research purposes unless you sign this consent form. By signing this consent form, you authorize the study doctor and his/her staff to use this information in conducting the study and to disclose and provide access to or copies of this information to the following:

- 1. Sponsor (Formation Biologics)
- 2. MedSource (contract research organization overseeing the study on the Sponsor's behalf), and other organizations working with the Sponsor to monitor the progress of the study or analyse the study data
- 3. (insert lab name) (local laboratory)
- 4. The U.S. Food and Drug Administration (FDA) or similar, national regulatory authorities
- 5. The (insert IRB/EC name) (IRB/EC) to ensure that patient safety and rights are protected

Access to this information is necessary to ensure that the study is being done correctly, and to collect and analyse data about the safety and effectiveness of the study medication.

You should know that once information is disclosed under this consent form to someone who is not a health care provider, the information is no longer protected. The Sponsor and those working with the

Sponsor on this study will only use and disclose your information as described in this consent form. If reports or articles are written about the study, your name will not appear on any report or publication.

You agree that, while the study is still in progress, you may not be given access to health information about you that is related to the study. While a request for access to health information can be denied, the study doctor and staff will consider whether it is medically appropriate under the circumstances to allow access. Your agreement that you may be denied access to your study-related health information during the study will not be used to deny you access to that information after the study is completed at all locations and study results are analysed.

You can only participate in the study if you authorize the use and disclosure of the information as described above. If you decide not to sign this consent form, you will not be enrolled in the study. If you sign this consent form and decide later to withdraw your consent, you will not be permitted to continue your participation in the study. Information collected up to the time that you withdraw your consent may continue to be used and disclosed as described above, but only as necessary to protect the integrity of the research study.

This authorization to use or disclose the information as described above is not time limited (that is, will not automatically expire).

You may decide not to sign this consent form, or you may revoke (withdraw) this authorization at any time. You can do this by giving written notice to your study doctor, informing him or her that you are revoking your consent to use and disclose your health information. The contact information for your study doctor is provided below.

| (insert name and telephone number of appropriate contact) |
|-----------------------------------------------------------|
| Study Doctor: |
| Address: |

#### **17.** YOUR RIGHTS AS A PARTICIPANT

Taking part in this study is voluntary. If you choose not to participate in this study, your care will not be affected. You may choose not to participate at any time during the study. Leaving the study will not affect your care.

We will tell you, in a timely manner, about significant new information that may affect your willingness to stay in this study.

You will be given a signed copy of this document. This consent form/authorization document does not

| have an exp | oiration date. | |
|---|---|---|
| | ther than the study doctor that your subjects, or research-related injury. | ou can call for information about the consent process, the rights ury is: |
| | (insert name and telephone nu | umber of appropriate contact) |
| | Contact Name: | |
| | Telephone Number: | |
| IRB or EC is questions co | s responsible for assuring that the<br>oncerning your rights in connec | tional Review Board (IRB) or an Ethics Committee (EC). The ne patients' safety, rights, and welfare are protected. If you have tion with this study, you can contact the IRB or EC. You may g address and telephone number. |
| | (insert name of IRB chairpers | son and/or name of IRB, address, and telephone number) |
| | IRB/EC contact: | |
| | Address: | |
| | Telephone Number | |
| 18. WH | HOM TO CONTACT IF YOU | HAVE QUESTIONS OR PROBLEMS |
| whether to ta | | eed more information about the study before you decide<br>em related to the study, you may contact the study doctor or<br>t page of this consent form. |
| - | ed on the first page of this conse | side effects during the study, call the study doctor at the ent form. If you are calling after hours or on a weekend, you |
| | (insert name and telephone nu | umber of appropriate contact) |
| | Contact Name: | |
| | Telephone Number: | |

# 19. CONSENT FOR STORED TUMOR TISSUE SCREENING FOR ELIGIBILITY AND BIOMARKER STUDIES

I understand that I am being asked to allow testing of my tumor at screening to determine if it is **positive** for the target of the study medication.

Because tumor tissue for testing is available from a prior biopsy or surgery I have undergone, I understand that I am being asked to consent to collection and testing of this tissue.

I also understand that I am being asked to consent to additional biomarker testing of my tumor for research purposes.

Based on study findings, and how I do on this study (if I participate), a request may be made for collection of additional stored tumor tissue after I begin treatment. I understand that agreement to collection of this additional tissue is **optional**.

# Patients asked to participate in Part 2:

| tumor is positive for the | ne target of the study m<br>tumor is not positive fo | red sample of my tumor to determine if my edication, and for other research purposes. I r the target of the study medication, I will not be |
|---|---|---|
| should such a request | be made. | tional stored sample of my tumor at a later date, at a stored sample of my tumor. |
| in the region of the permit | ission to concer and tec | it a stored sample of my tamor. |
| Signature of Patient | Date (mm/dd/yyyy) | Printed Name of Patient |
| Signature of Witness (relationship | Date (mm/dd/yyyy) | Printed Name of Witness |

Patients asked to participate in Part 2

to patient, if any)

#### 20. CONSENT FOR TUMOR BIOPSY FOR ELIGIBILITY AND BIOMARKER STUDIES

I understand that I am being asked to allow testing of my tumor at screening to determine if it is **positive** for the target of the study medication.

Because sufficient tumor tissue for testing is not available from a prior biopsy or surgery I have undergone, I understand that I am being asked to consent to a tumor biopsy to be performed

I also understand that I am being asked to consent to additional biomarker testing of my tumor for research purposes.

A tumor biopsy is a procedure in which a small sample of tumor is removed with a thin needle. Tumor biopsies will only be done if tumor tissue from the original site of the tumor, or from a site in your body where the tumor has spread, is thought to be easily accessible. Tumor sampling will only be attempted if a small sample can be taken with very little risk to you, and only if you agree to the procedure.

# Yes, I give permission to collect and test a biopsy sample of my tumor to determine if my tumor is positive for the target of the study medication, and for other for research purposes. I understand that if my tumor is not positive for the target of the study medication, I will not be eligible to participate in this study. No, I do not give permission to collect and test a biopsy sample of my tumor Signature of Patient Date (mm/dd/yyyy) Printed Name of Patient Printed Name of Witness

# 21. CONSENT FOR <u>OPTIONAL</u> COLLECTION OF TUMOR TISSUE FOR BIOMARKER STUDIES

I understand that I am being asked to allow additional testing of my tumor during the treatment portion of the study (after I have received study medication). I understand that this testing is optional, and if I refuse I may still participate in this study.

I understand that I am being asked to consent to the following:

- Release of a small portion of my tumor for testing, should I require surgery on an area of tumor while I am in the study
- A biopsy on an area of remaining tumor, should I have a response to study medication or a period of stable disease for more than 8 weeks
- A biopsy of my tumor, should study other findings suggest that more could be learned about the study medication if tumor tissue could be tested after dosing.

A tumor biopsy is a procedure in which a small sample of tumor is removed with a thin needle. Tumor biopsies will only be done if tumor tissue from the original site of the tumor, or from a site in your body where the tumor has spread, is thought to be easily accessible. Tumor sampling will only be attempted if a small sample can be taken with very little risk to you, and only if you agree to the procedure.

I also understand that I am being asked to consent to this additional **optional** biomarker testing of my tumor for research purposes.

# Patients asked to participate in Part 2

| | Yes, I give permission to collect and test a biopsy sample of my tumor for research purposes. understand that I may change my mind at a later time, if I choose to do so. | | |
|---|---|---|---|
| | No, I do not give permiss | ion to collect and test a b | piopsy sample of my tumor |
| Signa | ture of Patient | Date (mm/dd/yyyy) | Printed Name of Patient |
| _ | ture of Witness (relationship ient, if any) | Date (mm/dd/yyyy) | Printed Name of Witness |

Ι

Signature of Patient

#### 22. AGREEMENT TO CONSENT: PATIENT'S STATEMENT

The research project and treatment procedures associated with it have been fully explained to me. In addition, I have read the description of the clinical research study, or have had it translated into a language I understand. All experimental procedures have been identified and no guarantee has been given about the possible results. I have had the opportunity to ask questions concerning any and all aspects of the project and any procedures involved. I am aware that my primary doctor may be informed of my participation in this study, and that my primary doctor may be asked to provide information about my medical history. I am aware that participation is voluntary. I know that I may withdraw my consent at any time. I am aware that my decision not to take part, or to withdraw, will not restrict my access to health care services, and that I have not waived any of the legal rights that I would have if I were not a participant in a medical research study.

It has been explained to me that my personal data, including data relating to health or condition, and ethnic origin, may be used as described in this consent form, but that confidentiality of medical records concerning my involvement in this project will be maintained in an appropriate manner. When required by law, the records of this research may be reviewed by applicable government agencies, including the U.S. Food and Drug Administration (FDA) and Formation Biologics, or their representatives.

I, the undersigned, hereby voluntarily consent to participate as a patient in the above described research project. I will receive a copy of this consent for my records. I understand that if I have any questions concerning this research, or my rights in connection with the research, including if a research related injury occurs, I can contact the doctor(s) listed above. If I have questions concerning my rights in connection with the research, I can contact the Institutional Review Board or Ethics Committee, and that contact number has been provided to me.

Printed Name of Patient

Date (mm/dd/yyyy)

| Signature of Witness (relationship to patient, if any) | Date (mm/dd/yyyy) | Printed Name of Witness |
|---|---|---|
| I, the undersigned, certify that to t | he best of my knowled | INFORMED CONSENT DISCUSSION ge, the patient signing this consent form had the ds the nature, risks, and benefits of participation |
| Signature of Investigator (or Person Obtaining Consent) | Date (mm/dd/yyyy) | Printed Name of Person Obtaining Consent |